CLINICAL TRIAL: NCT06686836
Title: Efficacy of Platelet- and Leukocyte-rich Fibrin (L-PRF) in Reducing Healing Time in Sinus Lift Combined with Deproteinized Bovine Mineralized Bone (DBBM): Randomized Clinical Trial.
Brief Title: Efficacy of L-PRF Against Deproteinized Bovine Mineralized Bone (DBBM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Straumanngroup (Unknown); Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Juan Blanco Carrión, PhD, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECAELEV21; 2021-005374-26 (EudraCT Number)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Patients with Posterior Maxillary Atrophy and Need for Sinus Lift Surgery to Allow Implant Placement
Keywords: Posterior maxillary atrophy; Dental implants; Sinus lift; Bone grafting; Platelet-rich fibrin; Alveolar ridge augmentation; Bone regeneration; Bone substitutes
MeSH Terms: interventions — Bone Substitutes; Bio-Oss

STUDY DESIGN:
Intervention Model Description: The study compared two groups: one receiving DBBM alone (control) and the other receiving a combination of DBBM and an L-PRF block (test group).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Open sinus lift surgery using a bone substitute Bio-Oss®(Geistlich AG, Wolhusen, Switzerland) alone.
  Interventions: Procedure: Sinus lift augmentation with bone substitute (Bio-Oss)
- Test Group (Experimental): Open sinus lift surgery lift using Platelet- and leukocyte-rich fibrin (L-PRF) mixed with a bone substitute (Bio-Oss®(Geistlich AG, Wolhusen, Switzerland))
  Interventions: Procedure: Open sinus lift surgery lift using Platelet- and leukocyte-rich fibrin (L-PRF) mixed with a bone substitute (Bio-Oss®(Geistlich AG, Wolhusen, Switzerland)) - L-PRF Block

INTERVENTIONS:
Procedure: Sinus lift augmentation with bone substitute (Bio-Oss) — A maxillary sinus lift augmentation was performed with a lateral window approach that was filled with a bone substitute (Bio-Oss®) and covered with a collagen membrane (Bio-Guide®).At 4 months after sinus lift, a biopsy was taken and implants (Starumann®) were placed with submerged healing. After 6 months, the second surgical phase was performed and another biopsy was taken. The bone samples collected were analyzed histologically and histomorphometrically.
  Arms: Control Group
Procedure: Open sinus lift surgery lift using Platelet- and leukocyte-rich fibrin (L-PRF) mixed with a bone substitute (Bio-Oss®(Geistlich AG, Wolhusen, Switzerland)) - L-PRF Block — A maxillary sinus lift augmentation was performed with a lateral window approach that was filled using Platelet- and leukocyte-rich fibrin (L-PRF) mixed with a bone substitute (Bio-Oss®) and covered with a collagen membrane (Bio-Guide®) (L-PRF block).
  L-PRF block will be performed as described by Cortellini et al. 2018. L-PRF membranes are cut into small pieces and mixed with Bio-Oss® at a ratio of 2 membranes / 0.5 g biomaterial. Pieces of the block will be removed and compacted in the sinus cavity until it is filled.
  At 4 months after sinus lift, a biopsy was taken and implants (Starumann®) were placed with submerged healing. After 6 months, the second surgical phase was performed and another biopsy was taken. The bone samples collected were analyzed histologically and histomorphometrically.
  Arms: Test Group

SUMMARY:
Objective: The main objective of this study is to evaluate whether the use of L-PRF combined with deproteinized bovine mineralized bone (DBBM; BioOss, Geistlich Pharma®) reduces healing time, through histomorphometric analysis using bone biopsies after maxillary sinus elevation versus the use of deproteinized bovine mineralized bone (DBBM) alone.

Materials and methods: 24 patients with posterior maxillary atrophy (residual bone height <5mm without need for vertical regeneration) and need for sinus lift surgery to allow implant placement were treated ,12 DBBM (control group) 12 L-PRF block (Test group). At 4 months after sinus lift, a biopsy was taken and implants were placed with submerged healing. After 6 months, the second surgical phase was performed and another biopsy was taken. The bone samples collected were analyzed histologically and histomorphometrically. Patients received prosthetic restorations after 9 months and were followed up at 12 months. Volumetric changes were analyzed at 4 and 12 months.

DETAILED DESCRIPTION:
The study was a double-blind randomized controlled clinical trial (RCT), with a parallel design. Patients requiring an open sinus lift procedure before implant placement.

For the procedure it was use two types of filler, L-PRF block (test group) and DBBM alone (control group).

All patients were randomized and assigned to each of the study groups through a computer-generated randomization.

The primary outcome was percentage of new bone formed after treatment by histological and histomorphometric measurement of biopsies (%NeoformedBone=(Regenerated bone/total area)x100) at 4 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Presence of oral health (periodontally healthy or periodontitis treated), with a BoP <20% and PI <20%.
* Systemically healthy, with no disease that might contraindicate oral surgery.
* Non-smokers or smokers of <10 cig/day.
* Need to place implants in postero-superior sector with a residual bone height of < 5mm (no need for vertical regeneration).
* More than 3 months since tooth extraction in the treatment area.
* Absence of sinus pathology.

Exclusion Criteria:

* Patients who, due to systemic conditions, blood extraction is not possible.
* Medication that may interfere with bone metabolism (e.g. corticosteroids, bisphosphonates).
* History of radiotherapy.
* Pregnant and/or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Percentage of new bone formed | 4 and 6 months after treatment
  Measured by histological and histomorphometric analysis of biopsies at 4 and 6 months after sinus lift surgery

SECONDARY OUTCOMES:
Percentage of remaining material (%) | 4 and 6 months after treatment
  Measured by histology analysis at 4 and 6 months;
Volumetric changes of regenerated bone | baseline, 4 and 12 months after treatment
  Measured in millimeters according to CBCT at 4 and 12 months after maxillary sinus lift in apico-coronal and bucco-lingual orientation
Implant stability | 4 and 6 months after treatment
  Mesured ISQ (>65N) at the time of implant placement and in the second surgical phase before connecting the abutment to the implant).
Implant success | 12 months after treatment
  According to the criteria described by Misch,2008

CONTACTS AND LOCATIONS:
Locations (1):
- Department of periodontology, Faculty of Dentistry, University of Santiago de Compostela, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27783851/
- See also: Related Info — https://clinicaltrials.gov/fda-links
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16504861/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30690860/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21664828/